CLINICAL TRIAL: NCT04169646
Title: On-site Multi-component Intervention to Improve Productivity and Reduce the Economic and Personal Burden of Neck Pain in Swiss Office-Workers
Brief Title: Prevention and Intervention of Neck Pain in Swiss Office-Workers
Acronym: NEXpro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zurich University of Applied Sciences (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Principal Investigator, Markus Melloh, Principal Investigator, Zurich University of Applied Sciences
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 32003B_182389
Record Dates: First submitted 2019-11-13; First posted 2019-11-20 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Neck Pain; Headache; Musculoskeletal Diseases; Adherence, Patient; Absenteeism; Workplace; Health Promotion; Ergonomics; Efficiency; Presenteeism; Occupational Health; Surveys and Questionnaires; Adult; Exercise Therapy; Work Performance
Keywords: office-worker; neck-specific exercises; stepped wedge design; productivity
MeSH Terms: conditions — Neck Pain; Headache; Musculoskeletal Diseases; Patient Compliance | interventions — Health Promotion

STUDY DESIGN:
Intervention Model Description: This study is a stepped wedge cluster-randomized controlled trial.
Who Masked: Outcomes Assessor
Masking Description: A senior bio-statistician blinded to the identity of individuals will randomise clusters to a sequence within the period of data collection when clusters change from the control to the intervention condition (group 1 to 3).
  The outcome assessors of the physical examination will be blinded to group allocation and previous test results of the participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Other): Multi-component intervention
  Interventions: Other: Multi-component intervention
- Control (Other): Control
  Interventions: Other: Control

INTERVENTIONS:
Other: Multi-component intervention — Participants' workstation ergonomics will be assessed using an observation-based ergonomics assessment checklist for office-workers adapted to Swiss guidelines. Based on the initial assessment, best practice ergonomics will be applied individually using existing infrastructure. Participants will attend health promotion information group workshops for approximately one hour per week for 12 weeks. it. Participants will receive an individual progressive exercise programme aimed at conditioning the muscles of the neck and shoulder girdle. The exercises will be performed in groups (maximum of ten per group) at the workplace in a dedicated room, for approximately one hour (3x20 minutes) per week; once per week supervised by a physiotherapist, a human movement scientist, or a health scientist, and twice per week individually. Workshop session attendance will be recorded as an indication of adherence to health promotion. Adherence to neck exercises will be recorded with the Physitrack® app.
  Other Names: Workstation Ergonomics, Health promotion, Neck exercise, Adherence to intervention
  Arms: Intervention
Other: Control — No intervention takes place during the control phase.
  Arms: Control

SUMMARY:
This study is the first that investigates the impact of a multi-component intervention combining current evidence of effective interventions with an adherence app to assess the potential benefits on productivity, neck pain, and headache.

DETAILED DESCRIPTION:
Non-specific neck pain and headache are major economic and individual burdens in office-workers. The aim of this study is to investigate the effect of a multi-component intervention combining workstation ergonomics, health promotion information group workshops, neck exercises, and an app to enhance intervention adherence to assess possible reductions in the economic and individual burden of neck pain and headache in office workers.

This study is a stepped wedge cluster-randomized controlled trial. Eligible participants will be any office-worker aged 18-65 years from two Swiss organisations in the Canton of Zurich and Canton of Aargau, working more than 25 hours a week in predominantly sedentary office work and without serious health conditions of the neck. 120 voluntary participants will be assigned to 15 clusters which, at randomly selected time steps, switch from the control to the intervention group. The intervention will last 12 weeks and comprises workstation ergonomics, health promotion information group workshops, neck exercises and an adherence app. The primary outcome will be health-related productivity losses (presenteeism, absenteeism) using the Work Productivity and Activity Impairment Questionnaire. Secondary outcomes will include neck disability and pain. Physical and health outcomes (e.g. Neck Disability Index, muscle strength, and endurance), psychosocial outcomes (e.g. job-stress index, Fear-Avoidance Beliefs Questionnaire), workplace outcomes (e.g. workstation ergonomics), and individual outcomes (e.g. socio-demographic data, adherence to intervention) will be assessed. Measurements will take place at baseline, 4 months, 8 months, 12 months, 16 months, and 28 months after commencement. Data will be analysed on an 'intention to treat' basis and per protocol. Primary and secondary outcomes will be examined using linear mixed-effects models.

This study is the first that investigates the impact of a multi-component intervention combining current evidence of effective interventions with an adherence app to assess the potential benefits on productivity, neck pain, and headache. The outcomes will impact the individual, their workplace, as well as private and public policy by offering evidence for treatment and prevention of neck pain and headache in office-workers.

ELIGIBILITY:
Inclusion criteria:

* Swiss office-workers, who suffer from NP or want to take prevention of neck pain or headache
* 18-65 years old
* working more than 25 hours per week (0.6 full-time equivalent) in predominantly sedentary office work
* be able to communicate in German (written, spoken)
* have provided written informed consent

Exclusion criteria:

* previous trauma or injuries to the neck (NP grade 4)
* specific diagnosed pathologies (e.g., congenital cervical abnormalities, stenosis, fracture, radiculopathy)
* inflammatory condition (e.g., rheumatoid arthritis)
* any history of cervical spine surgery
* if exercise is contraindicated (e.g., medical advice, own beliefs)
* prolonged absence from work (more than four consecutive weeks) during the study intervention period
* pregnant women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Change in NP-related productivity loss | change from baseline at 16 months
  Change in NP-related productivity loss will be measured in percentages of the working time, using the Work Productivity and Activity Impairment Questionnaire for Specific Health Problem (WPAI German version) and converted into monetary units using individual earnings. Absenteeism is assessed by asking the participants about the number of hours missed because of NP as well as the number of hours they have actually worked. To assess presenteeism, the participants are asked to indicate on a 10-score scale how much the NP affected productivity while working, with 0 indicating no effect on productivity and 10 indicating total disability. Scoring rules of the developers of the questionnaire will then be used to obtain self-reported absenteeism and presenteeism expressed as impairment percentages. The monetary value for the lost productivity will be obtained for each individual by multiplying the impairment percentages by the individual gross wage.

SECONDARY OUTCOMES:
Neck pain | change from baseline at 16 months
  Neck pain intensity, occurence and frequency will be measured based on existing questionnaires (Standardised Nordic questionnaires for the analysis of musculoskeletal Symptoms; Neuromuscular assessment in Elderly Workers with and without work related) (open questions and numeric pain rating scale ranging from 0 to 10).
  neck/shoulder trouble).
Neck Disability Index | change from baseline at 16 months
  The German version of the Neck Disability Index (NDI) will be used to evaluate the extent to which NP interferes with vocational, recreational, social, and functional aspects of living. (score from 0 to 100)

OTHER OUTCOMES:
Physical activity level | baseline, after 4 months, after 8 months, after 12 months, after 16 months, after 28 months
  Short-form International Physical Activity Questionnaire (IPAQ German version) with data expressed as a continuous variable in metabolic equivalent of task (MET) min per week
Health related Quality of life | baseline, after 4 months, after 8 months, after 12 months, after 16 months, after 28 months
  The EuroQoL Five Dimension (ordinal scale) and EuroQoL visual analogue scale VAS (0-100 representing worst to best imaginable health state, respectively) will be used.
Job-Stress-Index | baseline, after 4 months, after 8 months, after 12 months, after 16 months, after 28 months
  The Job-Stress-Index provides the ratio between resources and work stressors. Normative statements (percentile ranks) will be given for representative groups of office-workers
Health beliefs | baseline, after 4 months, after 8 months, after 12 months, after 16 months, after 28 months
  Health beliefs will be assessed using three questions of the Fear-Avoidance Beliefs Questionnaire FABQ (dichotomous yes/no variable)
Psychosocial workplace factors | baseline, after 4 months, after 8 months, after 12 months, after 16 months, after 28 months
  Psychosocial workplace factors will be measured using a questionnaire (Copenhagen Psychosocial Questionnaire)
Workplace ergonomics | baseline, after 4 months, after 8 months, after 12 months, after 16 months, after 28 months
  observation-based ergonomics assessment checklist for office workers is adapted according to Swiss guidelines and used to assess the workplace ergonomics (dichotomous yes/no variable; score)
Work implementation | baseline, after 4 months, after 8 months, after 12 months, after 16 months, after 28 months
  a single question asking whether the participant felt their workplace culture supported the intervention (dichotomous yes/no variable).
Adherence to intervention | after 4 months, after 8 months, after 12 months, after 16 months, after 28 months
  neck and shoulder exercise performance and health promotion session attendance are documented. Next to this, participant's adherence to intervention (workplace ergonomics, exercises, health promotion) is asked using a self-reported scale (ordinal scale)
Participants' impression of change | after 4 months, after 8 months, after 12 months, after 16 months, after 28 months
  patients' global impression of change scale (PGIC) is used to reflect the participant's belief about the efficacy of intervention (numeric rating scale ranging from 0 to 10).
Care seeking | baseline, after 4 months, after 8 months, after 12 months, after 16 months, after 28 months
  Evaluated by two questions:
  * "Have you received healthcare services (e.g. doctor, physiotherapist, or other) because of work-related neck trouble in the past 12 months?" (yes/no; what)
  * "Have you required pharmaceutical medications due to neck trouble or headache in the last week?" (yes/no; what)
Breaks and Smartphone use | baseline, after 4 months, after 8 months, after 12 months, after 16 months, after 28 months
  three questions asking about the number of breaks during work, duration of each break (in minutes) and duration of daily smartphone use (in minutes)
Job satisfaction | baseline, after 4 months, after 8 months, after 12 months, after 16 months, after 28 months
  single item based on a 10-point numeric rating scale
Movement control | baseline, after 4 months, after 8 months, after 12 months, after 16 months, after 28 months
  Movement control dysfunction tests for the cervical spine (dichotomous, positive/negative)
Mobility of neck and head | baseline, after 4 months, after 8 months, after 12 months, after 16 months, after 28 months
  Mobility of the neck and head will be measured by an experienced and trained physiotherapist assessor using a CROM (range of motion, degree)
Muscle endurance | baseline, after 4 months, after 8 months, after 12 months, after 16 months, after 28 months
  Muscle endurance (time in seconds to task failure) of neck extensor and flexor muscles will be measured in a standardized testing position, either lying prone for neck extensors or supine for testing neck flexor muscles.
Muscle strength | baseline, after 4 months, after 8 months, after 12 months, after 16 months, after 28 months
  Muscle strength of neck extensor and flexor muscles and shoulder abductor muscles, in Newton peak force will be standardized measured with three repetitions and by using a handheld Dynamometer.
Pain pressure threshold | baseline, after 4 months, after 8 months, after 12 months, after 16 months, after 28 months
  Pain pressure threshold of the upper cervical spine (occiput, atlas) and of the trapezius muscle will be determined by using an Algometer.
Pain drawings | baseline, after 4 months, after 8 months, after 12 months, after 16 months, after 28 months
  Pain drawings: participants will be asked to complete their pain profile during the last week on two body charts (frontal and dorsal views) by using a pen. An operator will instruct the participants to shade their pain experience/complaints. The pain profile will include the aspects of pain extent (expressed as the percentage of the total body chart area where the pain will be reported), pain locations, pain intensity (using a numeric pain rating scale ranging from 0 to 10), location of the most painful spot, and pain intensity of the most painful spot (using a numeric pain rating scale ranging from 0 to 10).
Headache | baseline, after 4 months, after 8 months, after 12 months, after 16 months, after 28 months
  Headache will be measured using the questionnaire "headache impact test" (open questions and numeric pain rating scale ranging from 0 to 10).
Pre-existing headache conditions | baseline
  Pre-existing headache conditions will be screened for by an adapted headache screening questionnaire, based on validated German questionnaires (German Language Questionnaire for Screening for Migraine, Tension-Type Headache, and Trigeminal Autonomic Cephalgias; German-Language Self-Administered Headache Questionnaire; Der Rostocker Kopfschmerzfragen-Komplex)
Demographic information | baseline, (after 4 months, after 8 months, after 12 months, after 16 months, after 28 months)
  (self-reported) including employee's age (in years), sex, body-mass-index BMI (weight (kg) / height (m2)), duration of computer use/day (in minutes), occupation and income range (in CHF), working distance (in minutes, used transport system), general health conditions (diseases, nutrition, health literacy)

CONTACTS AND LOCATIONS:
Overall Officials: Markus Melloh, Prof, Principal Investigator — ZHAW School of Health Professions
Locations (2):
- Switzerland (2):
  - Kanton Aargau, Departement Bau, Verkehr und Umwelt, Aarau
  - ZHAW, Winterthur

IPD SHARING:
Plan to Share IPD: Yes
After the statistical analysis of this trial, the NEXpro team will make every endeavour to publish data in a journal (e.g. medical, health sciences). In particular, the following publications are planned: study protocol, primary outcome (productivity analysis), and several studies on the secondary and additional outcomes (e.g. neck pain analysis).
Supporting Information: Study Protocol
Time Frame: From June 2020 on (publication)
Access Criteria: Open access
URL: https://pubmed.ncbi.nlm.nih.gov/32560714/

REFERENCES:
- [Derived] Marchenko M, Domingues L, Barbero M, Cescon C, Falla D, Ernst MJ; NEXpro collaboration group. Headache, not neck pain, primarily influences the extent of pain in the neck region in symptomatic office workers. Cross-sectional and longitudinal evaluations. Physiother Theory Pract. 2025 Dec 12:1-11. doi: 10.1080/09593985.2025.2596179. Online ahead of print. PMID 41384674
- [Derived] Ernst MJ, Meichtry A, Luedtke K; NEXpro collaboration group; Falla D. Effects of neck-exercise and health promotion on headache outcomes in office workers: secondary analysis of the NEXpro stepped wedge cluster randomised controlled trial. J Headache Pain. 2025 Feb 12;26(1):30. doi: 10.1186/s10194-025-01963-y. PMID 39939850
- [Derived] Brunner B, Aegerter AM, Johnston V, Volken T, Deforth M, Sjogaard G, Elfering A, Melloh M; NEXpro Collaboration Group. Cost-utility and cost-benefit analysis of a multi-component intervention (NEXpro) for neck-related symptoms in Swiss office workers. BMC Public Health. 2025 Jan 15;25(1):160. doi: 10.1186/s12889-024-21103-6. PMID 39815202
- [Derived] Aegerter AM, Deforth M, Volken T, Johnston V, Luomajoki H, Dressel H, Dratva J, Ernst MJ, Distler O, Brunner B, Sjogaard G, Melloh M, Elfering A; NEXpro Collaboration Group. A Multi-component Intervention (NEXpro) Reduces Neck Pain-Related Work Productivity Loss: A Randomized Controlled Trial Among Swiss Office Workers. J Occup Rehabil. 2023 Jun;33(2):288-300. doi: 10.1007/s10926-022-10069-0. Epub 2022 Sep 27. PMID 36167936
- [Derived] Aegerter AM, Deforth M, Johnston V, Sjogaard G, Volken T, Luomajoki H, Dratva J, Dressel H, Distler O, Elfering A, Melloh M; NEXpro collaboration group. No evidence for an effect of working from home on neck pain and neck disability among Swiss office workers: Short-term impact of COVID-19. Eur Spine J. 2021 Jun;30(6):1699-1707. doi: 10.1007/s00586-021-06829-w. Epub 2021 Apr 4. PMID 33817763
- [Derived] Aegerter AM, Deforth M, Sjogaard G, Johnston V, Volken T, Luomajoki H, Dratva J, Dressel H, Distler O, Melloh M, Elfering A; NEXpro Collaboration Group. No Evidence for a Decrease in Physical Activity Among Swiss Office Workers During COVID-19: A Longitudinal Study. Front Psychol. 2021 Feb 11;12:620307. doi: 10.3389/fpsyg.2021.620307. eCollection 2021. PMID 33688857
- [Derived] Aegerter AM, Deforth M, Johnston V, Ernst MJ, Volken T, Luomajoki H, Brunner B, Dratva J, Sjogaard G, Elfering A, Melloh M; NEXpro collaboration group. On-site multi-component intervention to improve productivity and reduce the economic and personal burden of neck pain in Swiss office-workers (NEXpro): protocol for a cluster-randomized controlled trial. BMC Musculoskelet Disord. 2020 Jun 19;21(1):391. doi: 10.1186/s12891-020-03388-x. PMID 32560714